CLINICAL TRIAL: NCT00897377
Title: Treatment Strategy for Low-grade Gliomas
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Zhongping CHEN, Department of Neurosurgery, Sun Yat-sen University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YP2008009
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2009-05

CONDITIONS: Astrocytomas; Oligodendrogliomas; Oligoastrocytoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Total resection with early radiation (Experimental): Total resected LGGs treated with early radiation
  Interventions: Radiation: Radiation therapy
- Total resection without radiation (No Intervention): Total resected LGGs treated without radiation
- Residual LGGs with radiation (Experimental): Residual LGGs treated with early radiation
  Interventions: Radiation: Radiation therapy
- Residual LGGs with chemo (Experimental): Residual LGGS treated with temozolomide
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Radiation: Radiation therapy
  Arms: Residual LGGs with radiation; Total resection with early radiation
Drug: Temozolomide
  Arms: Residual LGGs with chemo

SUMMARY:
Although the prognosis of patients with low-grade glioma (LGG) is generally good, recurrence seems unavoidable in some patients because of the infiltrative growth of the tumors. How to treat LGGs is still under controversy. The role of radiation therapy and chemotherapy in the treatment of LGG need to be further investigated. The purpose of this study is the following:

1. to investigate the role of early radiation therapy in MRI-determined total resected LGGs;
2. to compare the efficacy of early radiation therapy and that of initial chemotherapy in the LGGs without total resection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed low-grade gliomas
* Karnofsky performance status of 60 or more

Exclusion Criteria:

* Previous history of radiation therapy or chemotherapy for gliomas
* Pregnant or breast feeding
* Diagnosis of another malignancy may exclude subject from study
* Evidence or history of bleeding diathesis
* Evidence or history of hypersensitivity to temozolomide

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-12

PRIMARY OUTCOMES:
Efficacy of early radiation therapy in MRI-determined total resected LGGs: evaluated as 5-year progression-free survival. | 10 years
Efficacy of early radiation therapy vs. initial chemotherapy with temozolomide in LGGs without total resection: evaluated as 5-year progression-free survival. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhongping Chen, M.D., Ph.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China